CLINICAL TRIAL: NCT01904851
Title: Multi-Center Registry Comparing Stent and Non-Stent Based Interventional Outcomes for Patients With Peripheral Arterial Disease
Brief Title: Multi-Center Registry for Peripheral Arterial Disease Interventions and Outcomes
Acronym: XLPAD
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STU 052012-093
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Stents; Registry; Angioplasty; Endovascular Procedures
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stent: The patient received one or more stents to the superficial femoral, popliteal, peroneal, anterior tibial, or posterior tibial arteries in AT LEAST one of the lesions treated during the course of the procedure.
- Non-Stent: The patient did not receive a stent to the superficial femoral, popliteal, peroneal, anterior tibial, or posterior tibial arteries in ANY of the lesions treated during the course of the procedure.

SUMMARY:
XLPAD is an observational study designed to evaluate the effectiveness and use of stent and non-stent based therapies among PAD patients. The study will create a registry that will include entry of procedural and clinical follow-up information into an online data collection software, REDCAP.Data available since Jan 1 2005 will be included in the registry, until 14,000 patients have been included. The primary objectives of this observational registry study are to:

1. Compare stent and non-stent based outcomes defined as a composite of symptom driven target vessel revascularization (TVR), unplanned surgical revascularization of the target limb and need for target limb amputation through 12 months post-index procedure (Primary efficacy endpoint)
2. Compare stent and non-stent based outcomes defined as a composite of causes such as: death, myocardial infarction (MI), stroke, peri-procedural complications, target vessel revascularization (TVR) and unplanned surgical revascularization/amputation of the target limb through 12 months (Primary safety endpoint)
3. Compare stent and non-stent based change in walking distance, Rutherford category and/or ankle- brachial index (ABI) at 12 months compared to baseline (Primary clinical improvement endpoint)

Approximately 14,000patients will be enrolled at approximately 60 sites worldwide. Enrollment in the observational study will be monitored in an effort to achieve at least 20% (and no more than 80%) of the population receiving stents as the initial treatment strategy. Follow-up visits by sites will be reported at 6 and 12 months after index procedure to collect data on treatment patterns and effectiveness, and outcomes. The follow-up procedures are not mandated by the registry protocol. Each site will be encouraged to enter follow-up information derived from clinically indicated follow-up visits. All events post-index procedure till the 7th month will be reported under the 6 month follow-up form and subsequent follow-up till the 13th month post-procedure will be entered on the 12 month follow-up form.

Patient management and treatment decisions are at the discretion of the care team per routine clinical practice. The procedural aspects (including selection of stent type or non-stent based treatments) and follow-up are not mandated by the registry and will be up to the discretion of the operator and/or based upon the practice dictated by the clinical care of the patient. Therefore the study poses minimal risk to the patient.

DETAILED DESCRIPTION:
Patients undergoing an endovascular intervention receiving either stents or percutaneous transluminal angioplasty (PTA) to the superficial femoral, popliteal, peroneal, anterior tibial, or posterior tibial arteries will be entered into this registry. Patients undergoing treatment of the external or common iliac arteries are not admissible to the registry, unless these arteries were treated in addition to one of the five aforementioned arteries. The registry will collect data in the form of patient background information, procedural data, and follow-up data from the patient's medical records. Data available since Jan 1 2005 will be included in the registry, until 14,000 patients have been included. The data will be entered into a software, REDCAP, that automatically provides data quality verification and processing.

Specifically, the data fields collected by the registry will be:

I) Background Information

1. Site, attending operator, and month-year of procedure
2. Patient height, weight, age, race, and sex
3. Rutherford claudication category, left and right ankle brachial index, ambulatory status, claudication free distance
4. Risk factors such as diabetes, hypertension, hyperlipidemia, and prior history of lower extremity percutaneous intervention
5. Patient comorbidities such as coronary artery disease, congestive heart failure, prior myocardial infarction, stroke, transient ischemic attack, chronic kidney disease, and other.

II) Lesion Characteristics (enter data for up to five lesions)

1. Access site relative to target limb, sheath size, target limb (left or right)
2. Target vessel: superficial femoral artery, popliteal artery, peroneal artery, anterior tibial artery, or posterior tibial artery
3. Which, if any, Iliac arteries were treated during procedure
4. Target lesion location (ostial, proximal, medial, distal), estimated vessel diameter, estimated vessel length
5. Lesion characteristics (heavily calcified, diffuse, thrombus, chronic total occlusion (CTO), in-stent restenosis, restenosis post balloon angioplasty, profunda femoris disease)
6. Planned revascularization strategy: stent or non-stent based

IIa) CTO Characteristics (Only required for CTO lesions)

1. Type of proximal and distal stumps, sidebranches present, collateral filling of distal vessel, tortuosity, prior attempt to cross CTO
2. Antegrade or retrograde crossing strategy, crossing technique, number of attempts
3. Crossing devices used, microcatheters used, sub-intimal re-entry devices used (if any), embolic protection device used

III) Intervention Details

1. Atherectomy device used (Cutting Balloon, TurboHawk, SilverHawk, Rotablator, Laser)
2. Pre and post-dilation balloon information (type, length, width, average atmospheric pressure, number of inflations)
3. Stent information (indication for stents, length, width, maximum pressure, overlapping with previous stents)
4. Aspiration/Thrombectomy used, thrombolytic therapy used
5. Percent change in stenosis and TIMI flows (before and after)

IV) Outcomes

1. Technical success (<30% residual stenosis), procedural success (<30% residual stenosis without complications), and case comments
2. Anti-coagulation used, medical therapy (plavix, aspirin, lipid lowering therapy, angiotensin receptor blocker, beta blocker, cilostazol, trental, insulin, oral hypoglycemics)
3. Duration of procedure, fluoroscopy (amount used, type, and time)
4. Any procedural complications

V) Follow-Up

1. Month and year of follow-up
2. Rutherford category, left and right ankle brachial index, claudication-free distance, ambulatory status, change in claudication (improved, same, or worsened)
3. Duplex ultrasound performed
4. Adverse events experienced (death, myocardial infarction, stroke, stent thrombosis, stent fracture, angiography, repeat endovascular intervention, surgical revascularization, amputation in target or non-target limb)

Follow-up data is recorded from clinical visits six and twelve months after the procedure. If the patient undergoes a repeat intervention on the target limb, a new record is created for the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Endovascular Intervention
* Treated Iliac, Common or Superficial Femoral, Popliteal, Peroneal, Anterior Tibial, or Posterior Tibial Arteries

Exclusion Criteria:

* Surgical Bypass

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed peripheral arterial disease who underwent endovascular intervention, and received either a stent or non-stent based treatment.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2013-01; Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Target Limb Revascularization | 12 months
  Target Lesion or Vessel Revascularization or Surgical Revascularization/Amputation of Target Limb

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — Baylor Research Institute
Locations (24):
- United States (24):
  - Arkansas Heart Institute, Little Rock, Arkansas
  - Denver VAMC, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Chicago, Illinois
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Mid West Cardiovascular Research Foundation, Davenport, Iowa
  - VA Boston Healthcare System, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - St. Louis University Medical Center, St Louis, Missouri
  - Carolina East Health System, New Bern, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Harrington Heart and Vascular Institute, University Hospitals, Cleveland, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Integris Heart Hospital, Oklahoma City, Oklahoma
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Seton Heart Institute/ UT Austin, Austin, Texas
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Christus Sphon Hospital Corpus Christi-Shoreline, Corpus Christi, Texas
  - North Texas Veteran Affairs Medical Center, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - El Paso Cardiovascular Care, El Paso, Texas
  - North Dallas Research Associates, McKinney, Texas
  - UT Health Sciences Center, San Antonio, Texas

REFERENCES:
- [Derived] Patel K, Liu Y, Etaee F, Patel C, Monteleone P, Patel M, Amer Alaiti M, Metzger C, Banerjee A, Minniefield N, Tejani I, Brilakis ES, Shishehbor MH, Banerjee S. Differences Between Patients With Intermittent Claudication and Critical Limb Ischemia Undergoing Endovascular Intervention: Insights From the Excellence in Peripheral Artery Disease Registry. Circ Cardiovasc Interv. 2021 Nov;14(11):e010635. doi: 10.1161/CIRCINTERVENTIONS.121.010635. Epub 2021 Oct 27. PMID 34706553
- [Derived] Armstrong EJ, Jeon-Slaughter H, Kahlon RS, Niazi KA, Shammas NW, Banerjee S. Comparative Outcomes of Supera Interwoven Nitinol vs Bare Nitinol Stents for the Treatment of Femoropopliteal Disease: Insights From the XLPAD Registry. J Endovasc Ther. 2020 Feb;27(1):60-65. doi: 10.1177/1526602819885652. Epub 2019 Nov 5. PMID 31686573
- [Derived] Kokkinidis DG, Jeon-Slaughter H, Khalili H, Brilakis ES, Shammas NW, Banerjee S, Armstrong EJ. Adjunctive stent use during endovascular intervention to the femoropopliteal artery with drug coated balloons: Insights from the XLPAD registry. Vasc Med. 2018 Aug;23(4):358-364. doi: 10.1177/1358863X18775593. Epub 2018 Jun 20. PMID 29923459
- [Derived] Shammas AN, Jeon-Slaughter H, Tsai S, Khalili H, Ali M, Xu H, Rodriguez G, Cawich I, Armstrong EJ, Brilakis ES, Banerjee S. Major Limb Outcomes Following Lower Extremity Endovascular Revascularization in Patients With and Without Diabetes Mellitus. J Endovasc Ther. 2017 Jun;24(3):376-382. doi: 10.1177/1526602817705135. Epub 2017 Apr 25. PMID 28440113
- [Derived] Banerjee S, Jeon-Slaughter H, Tsai S, Mohammad A, Foteh M, Abu-Fadel M, Gigliotti OS, Cawich I, Rodriguez G, Kumbhani D, Addo T, Luna M, Das TS, Prasad A, Armstrong EJ, Shammas NW, Brilakis ES. Comparative Assessment of Procedure Cost and Outcomes Between Guidewire and Crossing Device Strategies to Cross Peripheral Artery Chronic Total Occlusions. JACC Cardiovasc Interv. 2016 Nov 14;9(21):2243-2252. doi: 10.1016/j.jcin.2016.08.010. PMID 27832850
- [Derived] Banerjee S, Sarode K, Mohammad A, Gigliotti O, Baig MS, Tsai S, Shammas NW, Prasad A, Abu-Fadel M, Klein A, Armstrong EJ, Jeon-Slaughter H, Brilakis ES, Bhatt DL. Femoropopliteal Artery Stent Thrombosis: Report From the Excellence in Peripheral Artery Disease Registry. Circ Cardiovasc Interv. 2016 Feb;9(2):e002730. doi: 10.1161/CIRCINTERVENTIONS.115.002730. PMID 26839391
- [Derived] Banerjee S, Sarode K, Patel A, Mohammad A, Parikh R, Armstrong EJ, Tsai S, Shammas NW, Brilakis ES. Comparative Assessment of Guidewire and Microcatheter vs a Crossing Device-Based Strategy to Traverse Infrainguinal Peripheral Artery Chronic Total Occlusions. J Endovasc Ther. 2015 Aug;22(4):525-34. doi: 10.1177/1526602815587707. Epub 2015 May 18. PMID 25985785
- [Derived] Banerjee S, Thomas R, Sarode K, Mohammad A, Sethi S, Baig MS, Gigliotti OS, Ali MI, Klein A, Abu-Fadel MS, Shammas NW, Prasad A, Brilakis ES. Crossing of infrainguinal peripheral arterial chronic total occlusion with a blunt microdissection catheter. J Invasive Cardiol. 2014 Aug;26(8):363-9. PMID 25091095
- [Derived] Banerjee S, Sarode K, Das T, Hadidi O, Thomas R, Vinas A, Garg P, Mohammad A, Baig MS, Shammas NW, Brilakis ES. Endovascular treatment of infrainguinal chronic total occlusions using the TruePath device: features, handling, and 6-month outcomes. J Endovasc Ther. 2014 Apr;21(2):281-8. doi: 10.1583/13-4527R.1. PMID 24754288
- See also: XLPAD Registry Website — http://www.xlpad.org